CLINICAL TRIAL: NCT04105725
Title: A Mobile-based Behavioral Economic Intervention to Reduce Young Adult Alcohol Misuse
Brief Title: Balanced Lifestyle for Undergraduate Excellence - Mobile (Project BLUEM)
Acronym: BLUEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4324; 1F31AA026486-01A1 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-09-26 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Binge Drinking; Alcohol Drinking in College; Behavior, Drinking; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Binge Drinking; Alcohol Drinking in College; Drinking Behavior; Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI+Substance-Free Activity Session (Experimental): Two 50-minute text messaging sessions that discuss alcohol use and experiences related to alcohol use, as well as the individual's college, career, and personal goals. Additionally, there are 4 weeks of 20-30-minute booster text messaging sessions (once a week) that return to the individual's goals and progress.
  Interventions: Behavioral: Brief Motivational Intervention+Substance-Free Activity Session
- Alcohol + Nutrition Education Session (Active Comparator): Two 50-minute text messaging sessions the provide information on alcohol and nutrition. Additionally, there are 4 weeks of 20-30-minute booster text messaging sessions (once a week) that provide additional information and review previous information about alcohol use and nutrition.
  Interventions: Other: Alcohol + Nutrition Education Session

INTERVENTIONS:
Behavioral: Brief Motivational Intervention+Substance-Free Activity Session — A dialogue with the individual of their own experiences with alcohol use and related problems, as well as academic/career goals and personal interests.
  Other Names: BMI+SFAS; mBMI+SFAS; mobile BMI+SFAS
  Arms: BMI+Substance-Free Activity Session
Other: Alcohol + Nutrition Education Session — Education on alcohol, alcohol metabolism in the body, and alcohol overdose, as well as education on food groups and recommendations for a balanced diet.
  Other Names: A+NE; mA+NE; mobile A+NE
  Arms: Alcohol + Nutrition Education Session

SUMMARY:
The purpose of this study is to evaluate a text-message delivered approach for improving college adjustment and experience and reducing risky alcohol use in young adult college students. The study compares a text-message delivered brief motivational intervention for reducing alcohol use and increasing engagement in alcohol-free activities, to text-message delivered alcohol and nutrition education sessions. The investigators predict that individuals who receive the brief motivational intervention will report less alcohol use and fewer related problems 3 months following the intervention compared to those who receive the education sessions. The investigators also expect that these individuals will report greater engagement in alcohol-free activities compared to those who receive the education sessions.

DETAILED DESCRIPTION:
The proposed project will develop and empirically evaluate a mobile-based alcohol brief intervention and substance-free activity session. To do this, study personnel will develop and systematically evaluate an intervention that includes efficacious elements of brief alcohol interventions along with personalized feedback. Intervention elements will be delivered remotely via personalized web-based feedback and text-messages. The proposed project will evaluate the efficacy of the mobile-based brief alcohol intervention compared to mobile-based alcohol and nutrition education in the context of a randomized pilot trial.

This research will be divided into two stages: Stage 1, the screening stage, and Stage 2, the randomized pilot trial stage. During the screening stage, participants will be recruited and screened for eligibility to participate in Stage 2. The randomized controlled trial stage (stage 2) will test the feasibility and efficacy of a mobile-based BMI + SFAS in the context of a two-group experimental design. All students (N = 100) will complete a baseline assessment and will then be randomly assigned to either receive a mobile-based BMI + SFAS, or mobile-based alcohol and nutrition education. Each group will receive 4 weeks of booster contact (1 booster session per week) on material from their respective study condition. Outcomes will be assessed after the fourth booster session and at a 3-month follow-up.

Participants will complete a brief screening survey via the SONA system or through a secure web-link sent via email or posted in flyers to identify those students who might be eligible to participate in the study. In order to be contacted about the clinical trial, respondents will be asked to provide contact information. Ads and flyers will also include study contact information for interested respondents/participants to contact study staff directly and screen for eligibility.

If the participant meets eligibility criteria, the researcher will speak with the participant via phone call to explain the project procedures and confidentiality in more detail, and allow the participant the opportunity to ask any questions they may have about the study. Text messaging and email may also be used as methods to communicate with participants who meet the eligibility criteria and will be used as the primary method of communication if the student prefers. Participants will be informed that the study is designed to learn more about college students' lifestyle and health behaviors and that the study will involve random assignment to one of two treatment conditions, along with 4 booster sessions by text-message, a post-intervention survey immediately following the 4th booster session, and a survey follow-up three months after their last booster session. If the participant expresses interest in the study, the study administrator will invite them to participate in further phases of the study. If students do not meet the eligibility criteria at the time of screening, but indicate drinking in the past 6-months, they may be contacted later and re-screened via phone, text message or email and then enrolled if interested in the study. Eligible and interested individuals will remotely read and e-sign the consent form, provide contact information, and complete the initial baseline assessment via a secure web-link.

All self-report measures will be completed by the participant via a secure, web-based survey. Prior to completing baseline measures, participants will be provided with a consent form and will be informed of the study's purpose, risks, benefits, compensation, and all other pertinent study details. Participants will be provided with a phone number and email address should they have questions and will also be informed in the consent that they can discontinue the study at any time. If participants choose not to e-sign the consent form or decide not to participate in the study at any time, they will be provided with information about college student alcohol misuse on websites, hotlines, and local resources to learn more about their drinking if they are interested. The remote web-based assessment will last approximately 30 minutes. After completing the assessment, participants will be randomized to either a) the mobile-based BMI+SFAS (mBMI+SFAS); or b) mobile-based alcohol and nutrition education (mA+NE) (both described below). Immediately following the baseline assessment and random assignment, participants will take part in a 60-minute session of either the mobile BMI or mobile Alcohol Education. Later the same week, participants will take part in either one 60-minute session of the mobile SFAS or mobile Nutrition Education. The interventionist conducting the mobile BMI or Alcohol Education earlier in the week will also conduct the mobile SFAS or Nutrition Education, respectively, as well as all booster contact. A brief 3-item survey will be administered immediately following the mobile SFAS or Nutrition Education session that will solicit initial impressions and feedback on these respective sessions.

Booster contact will take place once a week for four weeks for approximately 20 minutes. Booster contact for the mBMI+SFAS group will also collect information on past week time allocation, level of discounting of future monetary rewards (delay discounting), and the subjective reward value of alcohol, which are associated with problematic alcohol use. Upon completion of the booster contact, participants will complete a 5-week assessment survey via secure web link. The post-intervention survey will collect information on the participants' experiences with the mobile-based interventions and will solicit feedback about the interventions. They will then be thanked for their participation and reminded of their 3-month follow-up appointment.

All participants will be asked to download on to their smartphone or personal computer a secure messaging web app called Babelnet (https://www.babelnet.com/en/). Babelnet is free to download and use, and study personnel will assist participants in the download and use of the app. Participants will be assigned a username that will be similar to their study identification number and a password that will be saved in a secure, password protected file only accessible to study personnel. In the event a participant has forgotten or lost their Babelnet login information, they may contact study personnel to retrieve it and log in securely. Messages sent through Babelnet are heavily encrypted by the app. However, study personnel will record (via screenshot or copy-and-paste) the text conversations to facilitate later communication and for intervention supervisory, as well as fidelity, purposes. These recordings will be saved on a secure server in a password protected shared drive that is accessible only to study personnel.

Three months post-booster completion, participants will be asked to remotely complete a web-based follow-up self-report assessment battery. The follow-up will assess the impact of the interventions on attitudes and behaviors toward alcohol use, as well as patterns of alcohol-related problems and drinking levels, and will last approximately 30 minutes.

After the 3-month assessment, participants will be given the option to complete any of the intervention sessions that they did not complete as a part of the study or to complete a session for a second time.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* Full-time college student
* Employed < or = 30 hours per week
* Report at least 2 past-month heavy drinking episodes (4 or more standard drinks for women and 5 or more standard drinks for men in one sitting/occasion)
* Own or have access to a smartphone, tablet, laptop, or desktop computer with Internet access
* Speak, read, and write in English

Exclusion Criteria:

* Currently in treatment for a substance use disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Soltis, M.S., Principal Investigator — The University of Memphis
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available for sharing with general research community 2 years after the grant end date on the Notice of Award (September 29, 2020), in order to provide study investigators with protected time to publish from the study data.
Time Frame: De-identified data will be made available September 30, 2022, which is two years after the project end date specified on the Notice of Award.
Access Criteria: De-identified data will be shared with qualified researchers with relevant expertise upon request for the purposes of conducting review papers or meta/integrated analyses.

RESULTS

PARTICIPANT FLOW:
Period: Primary Intervention
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 | 29
Completed | 37 | 26
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Mini-Session Week 1
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 36 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and Mini-Session Week 1) | 25 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and Mini-Session Week 1)
Not Completed | 1 | 1
Period: Mini-Session Week 2
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 34 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and Mini-Session Week 2) | 22 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and Mini-Session Week 2)
Not Completed | 3 | 4
Period: Mini-Session Week 3
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 34 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and Mini-Session Week 3) | 22 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and Mini-Session Week 3)
Not Completed | 3 | 4
Period: Mini-Session Week 4
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 35 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and Mini-Session Week 4) | 21 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and Mini-Session Week 4)
Not Completed | 2 | 5
Period: Post-Intervention Survey
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 33 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and the Post-Intervention Survey) | 18 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and the Post-Intervention Survey)
Not Completed | 4 | 8
Period: 3-Month Follow-up Survey
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Started | 37 (Number based on number completed both sessions of the BMI+Substance-Free Activity Session.) | 26 (Number based on number completed both sessions of the Alcohol + Nutrition Education Session.)
Completed | 33 (Number of participants who completed both sessions of the BMI+Substance-Free Activity Session and the 3-Month Follow-up Survey) | 22 (Number of participants who completed both sessions of the Alcohol + Nutrition Education and the 3-Month Follow-up Survey)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session | Total
Number analyzed (Participants) | 37 | 29 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.19 (1.63) | 19.66 (1.67) | 19.95 (1.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 34 | 24 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 22 | 17 | 39
  More than one race | 4 | 9 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 29 | 66
Daily Drinking Questionnaire [Mean (Standard Deviation); unit: typical drinks per week (past month)] | 11.86 (8.99) | 11.90 (8.57) | 11.88 (8.74)
Daily Drinking Questionnaire [Mean (Standard Deviation); unit: heavy drinking episodes (past month)] | 4.30 (3.66) | 4.59 (3.55) | 4.42 (3.59)
Brief Young Adult Alcohol Consequences Questionnaire [Mean (Standard Deviation); unit: # of consequences endorsed (past month)] | 8.57 (5.63) | 8.28 (5.69) | 8.44 (5.62)

OUTCOME MEASURES:

1. Primary Outcome: Daily Drinking Questionnaire
Description: Change in past-month typical weekly alcohol use
Time Frame: Baseline, 3-month follow-up
Measure: Mean (Standard Error); unit: drinks per week
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Number analyzed (Participants) | 31 | 20
drinks per week | 7.43 (0.85) | 8.11 (1.50)
Statistical Analysis 1: Comparison: Alcohol + Nutrition Education Session; Test type: Superiority; p < 0.05, negative binomial regression

2. Primary Outcome: Heavy Episodic (Binge) Drinking
Description: Change in past-month heavy drinking episodes
Time Frame: Baseline, 3-month follow-up
Measure: Mean (Standard Error); unit: past month heavy drinking episodes
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Number analyzed (Participants) | 31 | 20
past month heavy drinking episodes | 2.73 (0.54) | 4.04 (0.83)

3. Primary Outcome: Brief Young Adult Alcohol Consequences Questionnaire
Description: Change in past-month alcohol-related problems
Time Frame: Baseline, 3-month follow-up
Measure: Mean (Standard Error); unit: past month alcohol-related problems
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
Number analyzed (Participants) | 31 | 19
past month alcohol-related problems | 5.89 (0.89) | 5.13 (0.89)

4. Secondary Outcome: Adolescent Reinforcement Survey Schedule - Substance Use Version
Description: Change in substance-free reinforcement
Time Frame: Baseline, 5-week follow-up, 3-month follow-up
Reporting Status: Not Posted

5. Secondary Outcome: Monetary Choice Questionnaire
Description: Change in delay discounting
Time Frame: Baseline, 1-week follow-up, 2-week follow-up, 3-week follow-up, 4-week follow-up, 5-week follow-up, 3-month follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Alcohol Purchase Task
Description: Change in reinforcing efficacy (reward value) of alcohol
Time Frame: Baseline, 1-week follow-up, 2-week follow-up, 3-week follow-up, 4-week follow-up, 5-week follow-up, 3-month follow-up
Reporting Status: Not Posted

7. Secondary Outcome: Time Allocation
Description: Change in substance-free reinforcement
Time Frame: Baseline, 1-week follow-up, 2-week follow-up, 3-week follow-up, 4-week follow-up, 5-week follow-up, 3-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | BMI+Substance-Free Activity Session | Alcohol + Nutrition Education Session
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/29
Other Adverse Events (participants affected / at risk) | 0/37 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT04105725/Prot_SAP_ICF_000.pdf